CLINICAL TRIAL: NCT06283511
Title: Evaluation of the RESTART Survival Programme
Status: Not yet recruiting | Type: Observational
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IJB-RESTART
Record Dates: First submitted 2024-01-26; First posted 2024-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Invasive Breast Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: educational workshops — patient will be proposed to assist to educational workshops + the possibility to assist to a physical rehabilitation programme
  Other Names: physical rehabilitation programme

SUMMARY:
The RESTART survivorship programme has been implemented in the care pathway for patients with localised breast cancer since 2022. In this project, investigators are going to evaluate the satisfaction of patients taking part in the RESTART programme, as well as measuring changes in quality of life and health literacy after participation in the RESTART programme.

DETAILED DESCRIPTION:
Prospective longitudinal, single-centre, non-randomised study for patients who have completed acute treatment (surgery, radiotherapy, chemotherapy) for localised breast cancer within the last 3 months.

In this project, investigtors are going to evaluate the satisfaction of patients taking part in the RESTART programme, as well as measuring changes in quality of life and health literacy after participation in the RESTART programme.

The primary objective is to assess satisfaction with participation in the Restart programme and its various components.

Evaluation criteria associated with the primary objective:

Measurement of overall satisfaction and of the various components of the RESTART programme (Likert scale and open questions)

- Evaluation criteria associated with the secondary objective:

To measure before starting the RESTART programme and 1 and 12 months after the end of the programme:

* Patients' Quality of Life (QoL) (using the EORTC30 and BR23 questionnaires for breast cancer)
* Health literacy (via the HLQ questionnaire)
* Professional status
* Patients' physical activity level via the Global Physical Activity Questionnaire (GPAQ)
* Psychological distress, anxiety and depressive symptoms via the Generalized Anxiety Disorder - 7 (GAD-7) and Patient Health Questionnaire-9 (PHQ-9) questionnaires
* Fatigue (via the NRS)
* Patient sleep quality using the Pittsburgh Sleep Quality Index (PSQI) To measure the rate of participation in the programme via the proportion of patients who participated in relation to the number of patients operated on for breast cancer located in Bordet during the same period.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 at the time of signing the ICF
2. Minimum understanding of French
3. Signed study informed consent form obtained prior to any study-related procedure.
4. Participation in the RESTART programme
5. Patient with curative breast cancer (AJCC stage I-II-III)

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Refusal to participate in the RESTART programme
  2. Patients with AJCC stage IV breast cancer will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of satisfaction with participation in the Restart programme and its various components via Likert scale and open questions. | 1 month after end of programme and 12 months after end of the programme
  To assess the global satisfaction with participation in the Restart programme and its various components via the Likert Scale.

SECONDARY OUTCOMES:
assessment of quality of life | baseline - 1 month after end of programme - 12 months after end of programme
  To measure changes in quality of life via EORTC30 questionnaire
assessemnt of health literacy via HLQ questionnaire | baseline - 1 month after end of programme - 12 months after end of programme
  to mesure changes in health literacy via HLQ questionnaire
assessment of professional status | baseline - 1 month after end of programme- 12 months after end of programme
  to assess the number of patients who return to work via open question
assessment of level of physical activity | baseline - 1 month after end of programme- 12 months after end of programme
  to measure the changes in level of physical activity via the Global Physical Activity Questionnaire (GPAQ)
assessment of emotionnal distress | baseline - 1 month after end of programme- 12 months after end of programme
  to measure the changes in emotional distress via questionnaire "generalized Anxiety Disorder" (GAD-7)
assessment of the intensity of residual fatigue | baseline - 1 month after end of programme- 12 months after end of programme
  to measure the intensity of residual fatigue via NRS (0= no fatigue and 10 = worst fatigue)
assessment of sleep quality | baseline - 1 month after end of programme - 12 months after end of programme
  changes in sleep quality via Pittsburgh sleep Quality index (PSQI) before and after participation in the RESTART programme.
Measuring the rate of participation in the programme | baseline - 1 month after end of programme - 12 months after end of programme
  Measure the participation rate in the program via the proportion of patients who participated compared to the number of patients operated on for breast cancer located in Bordet during the same period.
assessment of quality of life | baseline - 1 month after end of programme - 12 months after end of programme
  To measure changes in quality of life via BR 23 questionnaire
assessment of emotionnal distress | baseline - 1 month after end of programme- 12 months after end of programme
  to measure the changes in emotional distress via questionnaire "Patient Health Questionnaire-9" (PHQ-9)

IPD SHARING:
Plan to Share IPD: No